CLINICAL TRIAL: NCT02380040
Title: Examination of Perfusion Index in Term and Preterm Newborns Through Plethismography
Brief Title: Plethismographic Perfusion Index in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 181/14
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Patent Ductus Arteriosus; Persistent Pulmonary Hypertension of the Newborn
MeSH Terms: conditions — Ductus Arteriosus, Patent; Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Term: Normal Term Newborn Intervention: PPG
  Interventions: Device: PPG
- Preterm: Preterm babies admitted to the NICU not suffering from the conditions to be studied Intervention: PPG
  Interventions: Device: PPG
- PDA: Patent Ductus Arteriosus Intervention: PPG
  Interventions: Device: PPG
- PPHN: Persistent Pulmonary Hypertension Intervention: PPG
  Interventions: Device: PPG

INTERVENTIONS:
Device: PPG — A PPG device will be applied to subjects in the right hand, left hand and one of the legs. Data will be recorded into a computer software

SUMMARY:
Photoplethismography will be measured and compared in newborns suffering from patent ductus arteriosus and normal controls.

DETAILED DESCRIPTION:
Newborn babies admitted to the NICU and well baby will be connected to a specially designed photoplethismograph (PPG). Right hand (pre ductal), and and one of the legs (postductal) values will be compared, based on the formula Delta amplitude of PPG / baseline absorption (perfusion index (PI)). Normal values will be defined in healthy term and preterm babies, and clinical conditions in which the PI is expected to change (Patent Ductus Artheriosus, Persistent pulmonary hypertension of the newborn)will be compared with these normal values.

ELIGIBILITY:
Inclusion Criteria:

* PDA, PPHN and Normal babies who underwent echocardiography

Exclusion Criteria:

* Other cardiac diseases

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and Preterm newborns admitted to the neonatology department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Perfusion Index | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Bromiker, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Ruben Bromiker, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nitzan I, Hammerman C, Fink D, Nitzan M, Koppel R, Bromiker R. The effect of patent ductus arteriosus on pre-ductal and post-ductal perfusion index in preterm neonates. Physiol Meas. 2018 Jul 20;39(7):075006. doi: 10.1088/1361-6579/aacf25. PMID 29943734